CLINICAL TRIAL: NCT04947137
Title: Development of a Normative Database for Rheumatoid Arthritis (RA) Imaging With Tc99m Tilmanocept
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-35
Record Dates: First submitted 2021-05-10; First posted 2021-07-01 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2022-03

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Healthy control; Tilmanocept
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, multicenter, single-dose study designed to develop a normative database of TUVjoint in HCs and to assess the feasibility of qualitative and quantitative SPECT/CT assessments in HCs and subjects with active RA. Subjects will be enrolled in 1 of 2 study arms with distinct study procedures in accordance with Arm-specific eligibility requirements.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects Free of Inflammatory Disease (Experimental): The first arm will be comprised of HCs who are deemed to be clinically free of inflammatory diseases, arthropathies, and/or arthroplasties and clinically free of joint pain for at least 28 days prior to the consent date.
  Interventions: Drug: Tc99m tilmanocept
- Healthy Controls and RA Subjects on Stable Therapy (Experimental): The second arm is comprised of [1] disease-free HCs and [2] clinically diagnosed RA subjects on stable treatment.
  Interventions: Drug: Tc99m tilmanocept

INTERVENTIONS:
Drug: Tc99m tilmanocept — Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
  Other Names: Lymphoseek

SUMMARY:
This study will establish a normative database of Tilmanocept Uptake Values (TUVjoint) in healthy controls age-matched to the RA population.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicenter, single-dose study designed to develop a normative database of TUVjoint in HCs and to assess the feasibility of qualitative and quantitative SPECT/CT assessments in HCs and subjects with active RA.

This study is stratified into 2 arms. Arm 1 is comprised of HCs and Arm 2 is comprised of HCs and clinically diagnosed RA subjects on stable treatment.

ELIGIBILITY:
Inclusion Criteria:

ALL SUBJECTS

1. The subject has provided written informed consent with HIPAA (Health Information Portability and Accountability Act) authorization before the initiation of any study-related procedures.
2. The subject has agreed to not engage in any diet, lifestyle, or medication changes until study completion.

   HEALTHY CONTROL SUBJECTS
3. The subject is 30 years of age or greater at the time of consent.
4. The subject is deemed to be clinically free of any inflammatory disease(s), autoimmune disease(s), or arthropathies and has not experienced joint pain for at least 28 days prior to the consent date.
5. The subject is not currently on anti-inflammatory drugs (including non-steroidal anti-inflammatory drugs [NSAIDs]) and has not taken any anti-inflammatories for at least 28 days prior to the consent date.
6. For all ongoing concomitant medications, the subject has maintained a stable dose for at least 28 days prior to the consent date.

CLINICALLY DIAGNOSED ACTIVE RA SUBJECTS

3. The subject is at least 18 years of age and was ≥ 18 years of age at the time of RA diagnosis.

4. The subject has moderate to severe RA as determined by the 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Classification Criteria (score of ≥ 6/10).

5. The subject has a 28-joint disease activity score (DAS28) of ≥ 3.2 (includes the Erythrocyte Sedimentation Rate [ESR] test and Visual Analog Scale [VAS]).

6. Subjects receiving traditional DMARDs must have been on therapy for ≥ 90 days and at a stable dose for ≥ 30 days prior to the imaging visit (Day 0). 7. If the subject is receiving bDMARD or janus kinase (JAK) inhibitor therapy, they have been at a stable dose > 60 days prior to the imaging visit (Day 0). 8. If the subject is receiving NSAIDs or oral corticosteroids, the dose has been stable for ≥ 28 days prior to the imaging visit (Day 0). The corticosteroid dose must be ≤ 10 mg/day of prednisone or an equivalent steroid dose.

Exclusion Criteria:

1. The subject is pregnant or lactating.
2. The subject size or weight is not compatible with imaging per the investigator.
3. The subject is currently receiving radiation therapy or chemotherapy or has received radiation therapy or chemotherapy in the past six months.
4. The subject has had a finger, hand, and/or wrist amputation or hand or wrist joint arthroplasty.
5. The subject has renal insufficiency as demonstrated by a glomerular filtration rate of < 60 mL/min.
6. The subject has hepatic insufficiency as demonstrated by ALT (alanine aminotransferase [SGPT]) or AST (aspartate aminotransferase [SGOT]) greater than 2 times the upper limit of normal.
7. The subject has any severe, acute, or chronic medical conditions and/or psychiatric conditions and/or laboratory abnormalities that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration that would deem the subject inappropriate for study participation or compromise the safety of the subject or the quality of the data.
8. The subject has any unstable medical illnesses, including hepatic, renal, gastroenterologic, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
9. The subject has a known allergy to or has had an adverse reaction to dextran exposure.
10. The subject has received an investigational product within 30 days prior to Tc 99m tilmanocept administration (Day 0).
11. The subject has received intra-articular corticosteroid injections ≤ 8 weeks prior to Tc 99m tilmanocept administration (Day 0).
12. The subject has received any radiopharmaceutical within 7 days or 10 half-lives prior to Tc 99m tilmanocept administration (Day 0).
13. Healthy Controls only: The subject has a positive rheumatoid factor and an elevated ESR or CRP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blue, MD, Study Director — Navidea Biopharmaceuticals
Locations (7):
- United States (7):
  - San Marcus Research Clinic, Miami Lakes, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Kettering Medical Center, Kettering, Ohio
  - Essential Medical Research, Tulsa, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Sun Research Institute, San Antonio, Texas
  - Tranquility Research, Webster, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Free of Inflammatory Disease: Arm 1 includes HCs who are deemed to be clinically free of inflammatory diseases, arthropathies, and/or arthroplasties and clinically free of joint pain for at least 28 days prior to the consent date.
  Tc 99m tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
- Healthy Controls and RA Subjects on Stable Therapy: Arm 2 includes [1] disease-free HCs and [2] clinically diagnosed RA subjects on stable treatment.
  Tc 99m tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
Period: Overall Study
Arm/Group | Subjects Free of Inflammatory Disease | Healthy Controls and RA Subjects on Stable Therapy
Started | 120 | 14
Completed | 120 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects were included in the ITD population. The PP population includes the ITD population without any major protocol deviations. There was one subject with a major protocol deviation. All subjects injected with Tc 99m tilmanocept are included in the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects Free of Inflammatory Disease | Healthy Controls and RA Subjects on Stable Therapy | Total
Number analyzed (Participants) | 120 | 14 | 134
Age, Continuous [Mean (Full Range); unit: years] | 54.9 [30 to 81] | 54.8 [34 to 77] | 54.9 [30 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 9 | 103
  Male | 26 | 5 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 73 | 0 | 73
  Not Hispanic or Latino | 47 | 14 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 109 | 13 | 122
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Normal Limits of TUVjoint in Healthy Subjects
Description: The normal limits of TUVjoint (on a per joint basis) in HC subjects, which are defined as the 5 and 95 percentiles of TUVjoint of bilateral joints (i.e., bilateral wrists, metacarpophalangeal joint [MCPs], proximal interphalangeal [PIPs]).
Time Frame: Up to 39 days
Population: Data not collected.
Groups:
- Primary Endpoint Arm 1 and 2. Secondary Endpoints Arm 1 and 2: Primary Endpoint Arm 1 The distribution of TUV joint in HC subjects were summarized with descriptive statistics: mean, standard deviation, n, minimum, maximum, and median per reader, joint, and view. The 5 and 95 percentiles will be estimated with quantile regression fitting an intercept as a fixed term. The lower and upper limits of normal TUV joint were determined using non-parametric confidence intervals and kernel density-based confidence intervals.
  Primary Endpoint Arm 2 Localization of tilmanocept in the hands and wrists were summarized with frequency counts and percentages by reader and joint.
  Secondary Endpoint Arm 1 Normal quantile plots were provided per joint and reader, along with the p-value for the Shapiro-Wilk test of normality.
  Secondary Endpoints Arm 2 SUV was calculated and summarized on both a per-joint and a total of all joints with summary statistics: mean, standard deviation, n, minimum, maximum, and median.
  The predictive value of planar scans for SPECT/CT qualitative findings was summarized per joint and reader with a crosstabulation and the uncertainty coefficients for row | column, column | row, and symmetric. The planar result was deemed to be "positive" (i.e., inflamed) if TUV joint > 95 percentile of the reader results for the same joint in Arm 1. Otherwise, the planar result was deemed to be "negative."
Arm/Group | Primary Endpoint Arm 1 and 2. Secondary Endpoints Arm 1 and 2
Number analyzed (Participants) | 0

2. Primary Outcome: Qualitative Evaluation of SPECT/CT for Tilmanocept Localization
Description: Presence/absence of tilmanocept localization in the hands and wrists will be summarized with frequency counts and percentages by reader and joint.
Time Frame: Up to 39 days
Population: Data not collected.
Arm/Group | Subjects Free of Inflammatory Disease | Healthy Controls and RA Subjects on Stable Therapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Normal Distribution of TUVjoint
Description: Applicability of the Normal (Gaussian) distribution to TUVjoint data as assessed by normal quantile plots provided per joint and reader and p-value for the Shapiro-Wilk test of Normality.
Time Frame: Up to 39 days
Population: Data not collected.
Arm/Group | Subjects Free of Inflammatory Disease | Healthy Controls and RA Subjects on Stable Therapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Quantitative Evaluation of SPECT/CT
Description: Determination of joint-specific standardized uptake value (SUV) from SPECT/CT imaging within synovial spaces of the bilateral hands and wrists in HCs and RA subjects.
Time Frame: Up to 39 days
Population: Data not collected.
Arm/Group | Subjects Free of Inflammatory Disease | Healthy Controls and RA Subjects on Stable Therapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Planar and SPECT/CT Comparison
Description: Assessment of the predictive value of planar scans for SPECT/CT scans.
Time Frame: Up to 39 days
Population: Data not collected.
Arm/Group | Subjects Free of Inflammatory Disease | Healthy Controls and RA Subjects on Stable Therapy
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Safety Objective: To Evaluate Safety Through the Examination of AE Incidence and Changes Over Time in Laboratory Tests, Vital Signs, and Physical Examination Findings.
Time Frame: Up to 39 days
Population: The safety population was evaluated, which is any subject injected with Tc 99m tilmanocept.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Free of Inflammatory Disease | Healthy Controls and RA Subjects on Stable Therapy
Number analyzed (Participants) | 120 | 14
Participants
  Adverse Events | 2 | 0
  Abnormal Clinical Lab Results | 1 | 0
  Abnormal Vital Signs | 2 | 0
  Abnormal Physical Examinations | 13 | 8

ADVERSE EVENTS:
Time Frame: Untoward medical events beginning on Visit 2 (Day 0) through Visit 3 (Day 5 ± 3) were recorded as adverse events.
Arm/Group | Subjects Free of Inflammatory Disease | Healthy Controls and RA Subjects on Stable Therapy
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/14
Other Adverse Events (participants affected / at risk) | 2/120 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Free of Inflammatory Disease (N=120) | Healthy Controls and RA Subjects on Stable Therapy (N=14)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Analysis of NAV3-35 trial data was halted prior to evaluation of the acquired planar and SPECT/CT images. Preliminary analysis of data from other trials indicated that the ability of Tc 99m tilmanocept imaging to predict response to anti-TNFα therapy in RA patients would not be sufficient for the product to be commercially viable. Therefore, further development of the product for this indication was halted. Note that all subjects had completed the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT04947137/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT04947137/SAP_001.pdf